CLINICAL TRIAL: NCT05618249
Title: Inventory of Inappropriate Prescriptions of Proton Pump Inhibitors (PPIs) in People Over 75 Years of Age When Taking Over a Patient Base in the SOULTZ Haut-Rhin Sector
Brief Title: Inventory of Inappropriate Prescriptions of Proton Pump Inhibitors (PPIs) in People Over 75 Years of Age
Acronym: Etaliepre-IPP
Status: Completed | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 7600
Record Dates: First submitted 2022-11-08; First posted 2022-11-16 (Actual); Last update posted 2023-12-15 (Actual); Status verified 2023-12

CONDITIONS: Peptic Ulcer Disease
Keywords: Peptic Ulcer Disease; Proton pump inhibitors; PPI
MeSH Terms: conditions — Peptic Ulcer

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study would have as a starting point the results of a request carried out by the Medical Service Grand Est of the Health Insurance aiming to evaluate the number of boxes of PPI reimbursed in town pharmacy, in patients over 75 years old in the Grand Est of France from 01/01/2018 to 31/12/2018.

It aims to highlight and quantify a possible inappropriate use of PPIs in private practice.

ELIGIBILITY:
Inclusion criteria:

* Patient over 75 years of age
* Patient with a PPI in the initial prescription
* Patient seen at least once between 01/01/2018 and 31/11/2019 in the general practice
* Patient who has not expressed his opposition, after information, to the reuse of his data for the purpose of this research.

Exclusion criteria:

* Patient having expressed his opposition to participate in the study
* Impossibility to give the patient informed information (difficulties in understanding the subject, ...)
* Patient under legal protection
* Patient under guardianship or curatorship
* Patient who is no longer followed up in the office following an entry into an institution (EHPAD)

Min Age: 75 Years | Sex: All
Age Groups: Older Adult
Study Population: Patient, over 75 years of age, with a PPI in the initial prescription
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-08-30 (Actual)

PRIMARY OUTCOMES:
Retrospective systematic analysis of patient prescriptions to identify possible inappropriate use of PPIs in private practice | Files analysed retrospectively from January 01, 2018 to December 31, 2019 will be examined

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Gériatrie - CHU de Strasbourg - France, Strasbourg, France